CLINICAL TRIAL: NCT01609881
Title: The Role of Prostaglandins in the Progression of Diabetic Retinopathy and the Therapeutic Efficacy of Topical Ketorolac (Acuvail)
Brief Title: The Role of Prostaglandins in the Progression of Diabetic Retinopathy
Acronym: Prostaglandin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to lack of funding
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Assistant Professor of Ophthalmology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12022
Record Dates: First submitted 2012-03-27; First posted 2012-06-01 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Inflammation
Keywords: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acuvail (Other): Acuvail as preventive for inflammation and possible decrease or prevent diabetic retinopathy. The study has four arms - diabetic ketorolac, diabetic control, normal eyes ketorolac, normal eyes control. patients are randomized to ketorolac or control.
  Interventions: Drug: Acuvail
- Placebo (Placebo Comparator): Placebo using artificial tear drops
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acuvail — Dosing of drug 3 days prior to surgery
  Other Names: Ketorolac 0.45%
  Arms: Acuvail
Other: Placebo — Artificial tears qid for 3 days preoperatively
  Other Names: tears
  Arms: Placebo

SUMMARY:
Objective of the research study:

1. To measure anterior chamber and vitreous ketorolac (Acuvail®) concentrations after topical administration in patients undergoing routine vitrectomy to determine the ability of the medication to penetrate into the anterior chamber and vitreous cavity, and to compare these levels to the IC50 for the cyclooxygenase-1 and -2 enzymes (COX-1 and COX-2)
2. To measure vitreous concentrations of prostaglandin subtypes (PGE, PGD, PGF) and other inflammatory mediators (Interleukin-1β [IL-1β], IL-6, IL-8, tumor necrosis factor [TNF]-α, VEGF) in both diabetic and nondiabetic patients undergoing vitrectomy
3. To determine if topical ketorolac (Acuvail®) can penetrate the anterior chamber and vitreous cavity sufficiently to decrease levels of intraocular inflammatory mediators that have been shown to be elevated in diabetic patients
4. To serve as a precursor to a 5-year longitudinal clinical trial to determine if chronically administered topical ketorolac (Acuvail®) can prevent, delay or slow diabetic retinopathy.

Research hypothesis

1. Ketorolac (Acuvail®) will penetrate the anterior chamber and vitreous cavity sufficiently to achieve levels above the IC50 for COX-1 and COX-2
2. Prostaglandin and other inflammatory mediator levels in the anterior chamber and vitreous cavity will be significantly higher among diabetic patients than nondiabetic controls
3. Acuvail® can significantly lower anterior chamber and vitreous cavity levels of prostaglandins and other inflammatory mediators in diabetic patients

DETAILED DESCRIPTION:
Patients who require vitrectomy for any indication and those meeting the inclusion/exclusion criteria will be included. Patients will be consented to participate in the study and for surgery.

Nondiabetic patients will be included in one of two groups. Twenty will receive topical ketorolac (Acuvail®) preoperatively for 3 days and then samples will be taken at the time of surgery. Twenty other patients will serve as controls for intraocular prostaglandin and cytokine levels (to be compared to diabetic patients). This group will not receive preoperative ketorolac (Acuvail®).

Diabetic patients will be included in one of two groups. Twenty patients will have intraocular prostaglandin and cytokine levels measured. Twenty other patients will be in the interventional group to determine if topical ketorolac (Acuvail®) can successfully lower intraocular prostaglandin and inflammatory cytokine levels.

In all cases, patients are undergoing vitreoretinal surgery as the surgical treatment of choice for their condition. For this study, undiluted samples will be drawn from the vitreous cavity and anterior chamber at the beginning of the vitrectomy. These samples will be stored, analyzed and frozen.

Samples will be tested for prostaglandin levels, in addition to other inflammatory cytokines, and ketorolac levels.

Three days of Acuvail® given four times per day was chosen, as previous studies have shown that one dose of ketorolac 0.4% achieves a peak aqueous concentration of 57.5 ng/mL,1 and that 12 doses over two days achieves an aqueous concentration of 1079 ng/mL.2 Both values are well above the IC50 for COX-1 (5.3 to 7.5 ng/mL) and COX-2 (33.9-45.2 ng/mL). The upper end of this dosing spectrum was chosen, as more doses and a longer duration of therapy is likely required to achieve sufficient vitreous levels to inhibit COX-1 and COX-2. This dosing regimen was also used in another clinical study that assessed ketorolac levels and prostaglandin levels in the vitreous cavity after topical administration four times a day for three days preoperatively.3

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years or older who present for vitrectomy surgery for any indication.
2. Diabetic and non-diabetic patients will be included.

Exclusion criteria:

1. Patients under the age of 18 years of age.
2. Pregnant women.
3. Patients with a history of vitrectomy surgery.
4. Current topical, periocular, intraocular or systemic corticosteroid use
5. Co-existent macular, retinovascular or ocular inflammatory disease (age-related macular degeneration, retinal venous occlusive disease, uveitis, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

PRIMARY OUTCOMES:
Vitreous and anterior chamber levels of prostaglandins, other cytokines, and Acuvail | 3 days
  Vitreous and anterior chamber levels of prostaglandins, other cytokines, and Acuvail

SECONDARY OUTCOMES:
Primary Outcome | 7 days
  The primary outcomes include drug and prostaglandin concentrations on the anterior chamber and vitreous.
Secondary Outcome | 14 days
  The secondary outcome will include cytokine levels in the vitreous.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt Eye Institute
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Schoenberger SD, Kim SJ, Shah R, Sheng J, Cherney E. Reduction of interleukin 8 and platelet-derived growth factor levels by topical ketorolac, 0.45%, in patients with diabetic retinopathy. JAMA Ophthalmol. 2014 Jan;132(1):32-7. doi: 10.1001/jamaophthalmol.2013.6203. PMID 24336915
- [Derived] Schoenberger SD, Kim SJ, Sheng J, Calcutt MW. Reduction of vitreous prostaglandin E2 levels after topical administration of ketorolac 0.45%. JAMA Ophthalmol. 2014 Feb;132(2):150-4. doi: 10.1001/jamaophthalmol.2013.5692. PMID 24264034
- [Derived] Schoenberger SD, Kim SJ, Sheng J, Rezaei KA, Lalezary M, Cherney E. Increased prostaglandin E2 (PGE2) levels in proliferative diabetic retinopathy, and correlation with VEGF and inflammatory cytokines. Invest Ophthalmol Vis Sci. 2012 Aug 27;53(9):5906-11. doi: 10.1167/iovs.12-10410. PMID 22871833